CLINICAL TRIAL: NCT01106066
Title: A Phase I/II Study of Neoadjuvant Chemoradiotherapy With S-1/ Oxaliplatin in Patients With Gastric Cancer
Brief Title: Phase I/II Study of Neoadjuvant Chemoradiotherapy With S-1/ Oxaliplatin in Patients With Gastric Cancer: Randomized Phase II Study of S-1/RT vs. S-1/Oxaliplatin/RT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruiting patients
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-06-013
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Phase I: To Determine the Maximum Tolerated Dose (MTD); Phase II: To Assess the Pathologic CR Rate and Feasibility Following Neoadjuvant Chemoradiation Therapy With S1/Oxaliplatin
MeSH Terms: interventions — Oxaliplatin; S 1 (combination); Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1/oxaliplatin/RT (Experimental): Radiotherapy + 4 dose levels of oxaliplatin/S-1
  Interventions: Drug: Oxaliplatin, S-1, radiotherapy

INTERVENTIONS:
Drug: Oxaliplatin, S-1, radiotherapy — Radiotherapy 4000cGy/20 fractions S-1 ( )mg/m2 po bid daily during radiotherapy Oxaliplatin at four dose levels (___mg/m2 iv weekly x 4 weeks)

SUMMARY:
To evaluate the efficacy of preoperative S-1/oxaliplatin/RT in locally advanced gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years

  * Patients with localized, histologically confirmed gastric or gastroesophageal adenocarcinoma ③ Localized gastric cancer of clinical stage (T2N(+), T3/T4)

    * ECOG performance status of 0 to 1 ⑤ Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; total bilirubin ≤1.5 UNL; AST and/or ALT < 5 UNL; creatinine clearance ≥ 50mL/min ⑥ Written informed consent form

Exclusion Criteria:

* T1 (regardless of N stage), T2N0

  * M1 ③ Peritoneal seeding ④ Uncontrolled medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
MTD/pathologic CR | at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Cancer Center, Seoul, South Korea